CLINICAL TRIAL: NCT00381550
Title: Phase II Trial of Triapine (NSC #663249, 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbone) Plus Fludarabine (NSC #312887, Fludarabine Monophosphate) in Adults With Aggressive Myeloproliferative Disorders (MPDs) Including Chronic Myelomonocytic Leukemia (CMML) and Chronic Myelogenous Leukemia in Accelerated Phase (CML-AP) or Blast Crisis (CML-BC)
Brief Title: 3-AP and Fludarabine in Treating Patients With Myeloproliferative Disorders, Chronic Myelomonocytic Leukemia, or Accelerated Phase or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00209; NCI-2009-00209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J0638 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 7704 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2014-05-21 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Essential Thrombocythemia; Philadelphia Chromosome Negative Chronic Myelogenous Leukemia; Polycythemia Vera; Primary Myelofibrosis; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — fludarabine phosphate; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive 3-AP (Triapine®) IV over 4 hours followed by fludarabine phosphate IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fludarabine phosphate; Drug: triapine; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Procedure: laboratory biomarker analysis — Correlative study

SUMMARY:
This phase II trial is studying how well giving 3-AP together with fludarabine works in treating patients with myeloproliferative disorders (MPD), chronic myelomonocytic leukemia (CMML), or accelerated phase or blastic phase chronic myelogenous leukemia. Drugs used in chemotherapy, such as 3-AP and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. 3-AP may help fludarabine work better by making cancer cells more sensitive to the drug. 3-AP and fludarabine may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving 3-AP together with fludarabine may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of 3-AP (Triapine®) followed by fludarabine phosphate in patients with myeloproliferative disorders or chronic myelomonocytic leukemia in aggressive phase or transformation or chronic myelogenous leukemia in accelerated phase or blast crisis.

II. Determine the toxicity of this regimen in these patients. III. Determine, preliminarily, the effect of this regimen on circulating leukemic cell genetics in these patients.

Outline: This is an open-label study.

Patients receive 3-AP (Triapine®) IV over 4 hours followed by fludarabine phosphate IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow and/or peripheral blood collection at baseline and periodically during study treatment for molecular analysis of Janus kinase 2 (JAK2) mutations, GATA-1 mutations, and expression of the death-inducer-obliterator (Dido) genes on chromosome 20q.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Criteria:

* Not pregnant or nursing
* Histopathologically confirmed diagnosis of 1 of the following:

  * Myeloproliferative disorders (MPDs) in aggressive phase or transformation
  * CML in accelerated phase or blast crisis
  * Chronic myelomonocytic leukemia in aggressive phase (5-19% bone marrow blasts) or transformation (> 20% bone marrow blasts)
* Myeloproliferative disorders (MPDs) in aggressive phase or transformation, including the following:

  * Polycythemia vera (PV)
  * Essential thrombocythemia (ET)
  * Myelofibrosis with myeloid metaplasia
  * Hypereosinophilic syndrome
  * Atypical (Philadelphia chromosome negative) chronic myelogenous leukemia (Ph- CML)
* Patients with aggressive phase MPD (PV, ET, or Ph- CML) must meet ≥ 1 of the following criteria:

  * Marrow blasts > 5%
  * Peripheral blood blasts plus progranulocytes > 10%
  * New onset or increasing myelofibrosis
  * New onset or > 25% increase in hepatomegaly or splenomegaly
  * New onset constitutional symptoms (fever, weight loss, splenic pain, bone pain)
* Multilineage bone marrow failure
* Ineligible for established curative regimens, including stem cell transplantation
* ECOG performance status 0-2
* Negative pregnancy test
* Fertile patients must use effective contraception
* No chronic toxicity from prior chemotherapy > grade 1
* No history of severe coronary artery disease
* Creatinine normal OR creatinine clearance >= 60 mL/min
* AST and ALT =< 2.5 times normal
* Bilirubin =< 2.0 mg/dL unless due to leukemia, Gilbert's syndrome, or hemolysis
* No arrhythmias (other than atrial flutter or fibrillation) requiring medication
* No uncontrolled congestive heart failure
* No dyspnea at rest or with minimal exertion
* No severe pulmonary disease requiring supplemental oxygen
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to 3-AP (Triapine®) and/or fludarabine phosphate
* No other life-threatening illness
* No history of mental deficits and/or psychiatric illness that would preclude study compliance
* No more than 4 prior induction regimens (3 cytotoxic chemotherapy regimens)
* At least 3 weeks since prior myelosuppressive cytotoxic agents (6 weeks for mitomycin C or nitrosoureas) and recovered
* At least 1 week since prior nonmyelosuppressive treatment
* At least 48 hours since prior noncytotoxic agents for peripheral blood leukemic cell count control, including but not limited to the following:

  * Hydroxyurea
  * Imatinib mesylate
  * Interferon
  * Mercaptopurine
  * Cyclophosphamide
* At least 2 weeks since prior and no concurrent radiotherapy to treat cancer
* At least 1 week since prior biologic therapy, including hematopoietic growth factors (e.g., epoetin alfa, darbepoetin alfa, filgrastim [G-CSF], sargramostim [GM-CSF], interleukin-3, or interleukin-11)
* No other concurrent chemotherapy to treat cancer
* No concurrent immunotherapy to treat cancer
* No known glucose-6-phosphate dehydrogenase [G6PD) deficiency (G6PD screening required for high-risk groups (i.e., patients of African, Asian, or Mediterranean origin/ancestry)]
* No active heart disease
* No concurrent myeloid growth factors
* No active uncontrolled infection (Infections under active treatment and controlled with antibiotics are allowed)
* No chronic hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Zeidner JF, Karp JE, Blackford AL, Smith BD, Gojo I, Gore SD, Levis MJ, Carraway HE, Greer JM, Ivy SP, Pratz KW, McDevitt MA. A phase II trial of sequential ribonucleotide reductase inhibition in aggressive myeloproliferative neoplasms. Haematologica. 2014 Apr;99(4):672-8. doi: 10.3324/haematol.2013.097246. Epub 2013 Dec 20. PMID 24362550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient's presenting for treatment of a myeloproliferative disease were considered for participation.
Pre-assignment Details: Once patient consented to treatment, treatment began shortly there after.
Groups:
- Triapine and Fludarabine Phosphate: Patients receive 3-AP (Triapine®) IV over 4 hours followed by fludarabine phosphate IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Triapine and Fludarabine Phosphate
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Response Rate Including Complete Response, Partial Response, and Hematological Improvement Assessed by Blood Cell Counts, Number of Blasts in Bone Marrow, and Clinical Evaluation
Description: Bone marrow aspiration and biopsies were performed prior to treatment, during week 3 of the first cycle, at the time of hematologic recovery from all cycles of therapy (defined as neutrophil count >500/mm3 and platelets >20,000/mm3 independently of transfusion), or at any time that leukemia regrowth was suspected. The overall response rate was defined as complete remission, partial remission, or hematologic improvement, lasting for ≥30 days. Given the different subsets of diseases, standardized response criteria were used for CMML (the Myelodysplastic Syndrome International Working Group criteria),33 CMML transforming to acute myeloid leukemia (standard AML response criteria) , accelerated MPN (Giles et al.), and transformation of MPN to secondary AML (Mascarenhas et al.).
Time Frame: Up to 4 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 35
participants | 18

2. Primary Outcome: Incidence of Grade 3 or 4 Drug-related Non-hematologic Toxicity as Assessed by NCI CTCAE v3.0
Time Frame: Up to 4 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 35
participants | 35

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 18/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=35)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2)
Tumor Lysis syndrome (Metabolism and nutrition disorders) | 3 (3)
Infections (Infections and infestations) | 7 (7)
Kidney injury (Investigations) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=35)
Acidosis (Metabolism and nutrition disorders) | 10 (10)
Allergic reaction (General disorders) | 5 (5)
Anaphylaxis (General disorders) | 2 (2)
Elevated bilirubin (Metabolism and nutrition disorders) | 14 (14)
Elevated creatinine (Metabolism and nutrition disorders) | 8 (8)
Fever (General disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less